CLINICAL TRIAL: NCT00001672
Title: Language Localization Using Repetitive Transcranial Magnetic Stimulation (rTMS) in Patients With Epilepsy
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970175; 97-N-0175
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-08

CONDITIONS: Epilepsy, Temporal Lobe
Keywords: Brain Mapping; Cognition; Noninvasive; Temporal Lobe; Visual Naming
MeSH Terms: conditions — Epilepsy, Temporal Lobe

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) may be able to provide a moderately detailed localization of language functions in the brain. We propose to test the ability of rTMS to locate the substrate of visual naming to a limited area of the temporal lobe in patients with temporal lobe epilepsy before and after surgical resections. The study is expected to yield information on the organization of language in the temporal lobes and how unilateral temporal lobe lesions and lobectomy cause relocation of language mechanisms in the lesioned and in the other hemisphere. It will also be a preliminary step in the development of a clinically useful procedure for locating critical language areas in potential surgical candidates.

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation (rTMS) may be able to provide a moderately detailed localization of language functions in the brain. We propose to test the ability of rTMS to locate the substrate of visual naming to a limited area of the temporal lobe in patients with temporal lobe epilepsy before and after surgical resections. The study is expected to yield information on the organization of language in the temporal lobes and how unilateral temporal lobe lesions and lobectomy cause relocation of language mechanisms in the lesioned and in the other hemisphere. It will also be a preliminary step in the development of a clinically useful procedure for locating critical language areas in potential surgical candidates.

ELIGIBILITY:
Patients will be drawn from among those referred to the NINDS Epilepsy Research Branch.

No patients with evidence for a progressive neurological disorder.

No subjects with metal hardware in the cranial cavity, cardiac pacemakers, indwelling medication pumps, cochlear implants, intracardiac lines, significant intracranial masses or evidence of increased intracranial pressure.

Women must not be pregnant.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 1997-09; Study Completion 2000-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Claus D, Weis M, Treig T, Lang C, Eichhorn KF, Sembach O. Influence of repetitive magnetic stimuli on verbal comprehension. J Neurol. 1993;240(3):149-50. doi: 10.1007/BF00857519. PMID 8482986
- [Background] Desmond JE, Sum JM, Wagner AD, Demb JB, Shear PK, Glover GH, Gabrieli JD, Morrell MJ. Functional MRI measurement of language lateralization in Wada-tested patients. Brain. 1995 Dec;118 ( Pt 6):1411-9. doi: 10.1093/brain/118.6.1411. PMID 8595473
- [Background] Epstein CM, Lah JJ, Meador K, Weissman JD, Gaitan LE, Dihenia B. Optimum stimulus parameters for lateralized suppression of speech with magnetic brain stimulation. Neurology. 1996 Dec;47(6):1590-3. doi: 10.1212/wnl.47.6.1590. PMID 8960755